CLINICAL TRIAL: NCT06676384
Title: Randomized Embedded Adaptive Platform Clinical Trial in South Asian Kidney Biopsy-Proven Primary IgA Nephropathy: Multi-center, Multi-arm and Multi-stage
Brief Title: Which of the Commonly Available and Approved Drugs in Addition to Standard of Care Can Significantly Improve the Slope of Estimated Glomerular Filtration Rate at Two Years When Compared to Standard of Care Alone in South-Asian Kidney Biopsy-proven Adult (≥18 Years) Primary IgA Nephropathy?
Acronym: IA-GRACE-IgANT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Christian Medical College, Vellore, India (Other)
Collaborators: Medical Research Council (Other Government); India Alliance (Unknown)
Responsible Party: Principal Investigator, Suceena Alexander, Professor and HoU (Nephrology Unit III), Christian Medical College, Vellore, India
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IA/CPHS/22/1/506541; IA/CPHS/22/1/506541 (Other Grant/Funding Number: DBT/WELLCOME TRUST INDIA ALLIANCE); 15811[INTERVEN] dated 25.10.23 (Other: CMC SILVER IRB & ETHICS COMMITTEE); CTRI/2024/11/076794 (Other: ICMR)
Record Dates: First submitted 2024-10-26; First posted 2024-11-06 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: IgA Nephropathy; Renal Insufficiency, Chronic; IgA Vasculitis; IGA Glomerulonephritis
Keywords: Platform Trial; Randomised Embedded Trial; MAMS Trial; IgA Nephropathy; Chronic kidney disease; Glomerulonephritis; IgA Vasculitis; Single blind; Treatment
MeSH Terms: conditions — Glomerulonephritis, IGA; Renal Insufficiency, Chronic; IgA Vasculitis; Glomerulonephritis | interventions — Prednisolone; Mycophenolic Acid; Hydroxychloroquine; Angiotensin Receptor Antagonists

STUDY DESIGN:
Intervention Model Description: This is a Phase 4 multi-arm, multi-stage (MAMS) platform trial. It is a multicenter, randomised, single-blind (outcome assessor), active comparator trial. The participants will be randomised 1:1 to the comparator and each of the four interventional arms. The sample size of 585 participants is for five arms, including the active comparator. The sixth arm may begin after the planned interim analysis conditional to the availability of the generic drug in the Indian market and will recruit additional 117 participants with concurrent comparator arm.
Who Masked: Outcomes Assessor
Masking Description: The statistician/ outcome assessor will be blinded to the drug allocation and use coded data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Standard of Care (SoC) (Active Comparator): This intervention arm will start with the randomisation of the first participant.
  Interventions: Drug: SoC defined as maximal labelled or tolerated dose of angiotensin-converting enzyme inhibitor/ angiotensin receptor blocker (ACEi/ARB) & steady dose of sodium-glucose cotransporter-2 inhibitor (SGLT2i)
- SoC and Oral prednisolone (Experimental): This intervention arm will start with randomisation of the first participant.
  Interventions: Drug: Oral prednisolone and SoC
- SoC and Gut-directed budesonide (Experimental): This intervention arm will start with the randomisation of the first participant.
  Interventions: Drug: Gut-directed budesonide and SoC
- SoC and Mycophenolate mofetil (MMF) (Experimental): This intervention arm will start with the randomisation of the first participant.
  Interventions: Drug: Mycophenolate mofetil (MMF) and SoC
- SoC and Hydroxychloroquine (Experimental): This intervention arm will start with the randomisation of the first participant.
  Interventions: Drug: Hydroxychloroquine and SoC
- SoC and Non-steroidal mineralocorticoid receptor antagonist (Experimental): The sixth arm may begin after the planned interim analysis conditional to the availability of the generic drug in the Indian market and will recruit an additional 117 participants with a concurrent comparator arm.
  Interventions: Drug: Non-steroidal mineralocorticoid receptor antagonist and SoC

INTERVENTIONS:
Drug: Oral prednisolone and SoC — Oral prednisolone 0.5 mg/kg per day (maximum, 40 mg/day) for two months, followed by dose tapering by 5mg per day each month for six to nine months. All participants in this arm will receive SoC and oral cotrimoxazole prophylaxis.
  Other Names: Wysolone® by Pfizer Ltd.
  Arms: SoC and Oral prednisolone
Drug: Gut-directed budesonide and SoC — Gut-directed Budesonide 12 mg once daily for nine months and tapered to 9mg once daily for the next three months, 6mg once daily for the next three months and 3mg once daily for the next three months and stopped (total 18 months). All participants in this arm will receive SoC.
  Other Names: IgANEF® by MediART Life Sciences Pvt. Ltd.
  Arms: SoC and Gut-directed budesonide
Drug: Mycophenolate mofetil (MMF) and SoC — Mycophenolate mofetil (MMF) 1.5g/ day for twelve months, followed by 1g/ day for six months (total 18 months). All participants in this arm will receive SoC.
  Other Names: Mycept® by Panacea Biotec Ltd.
  Arms: SoC and Mycophenolate mofetil (MMF)
Drug: Hydroxychloroquine and SoC — Hydroxychloroquine (HCQ) 6.5 mg/kg/day (maximum 400 mg daily) for 24 months. All participants in this arm will receive SoC.
  Other Names: Ipca HCQ® by IPCA Laboratories Ltd.
  Arms: SoC and Hydroxychloroquine
Drug: Non-steroidal mineralocorticoid receptor antagonist and SoC — Generic drug not available currently. All participants in this arm will receive SoC.
  Arms: SoC and Non-steroidal mineralocorticoid receptor antagonist
Drug: SoC defined as maximal labelled or tolerated dose of angiotensin-converting enzyme inhibitor/ angiotensin receptor blocker (ACEi/ARB) & steady dose of sodium-glucose cotransporter-2 inhibitor (SGLT2i) — Maximal labelled or tolerated dose of ACEi/ ARB and a steady dose of SGLT2i (10mg/d of dapagliflozin).
  Other Names: Dapmed® by Medgenix Pharma India Pvt. Ltd.
  Arms: Standard of Care (SoC)

SUMMARY:
Global Burden of Diseases ranks chronic kidney disease (CKD) as the 12th leading cause of death, with an estimated 20% increase from 2010 to 2019. India is the most populous country in South Asia, with one-fourth of the global population. CKD prevalence has reached epidemic proportions in South Asia, with 1 in 7 adults affected by it. Glomerular diseases are the most common cause of CKD after diabetes and hypertension. IgAN is the most common primary glomerular disease in adults. In the Caucasian and East Asian populations, IgAN results in end-stage kidney disease (ESKD) in 15-20% of patients within 15-20 years after the first clinical presentation.

Our first prospective observational (GRACE-IgANI) cohort since 2015 showed that South Asians have severe and progressive IgAN, with 39% having a rapid fall in eGFR, 25% having non-remission of proteinuria, and 36% reaching an adverse kidney outcome at three years. Our group has shown that South Asian ethnicity is associated with a severe phenotype, rapid progression, and significant ethnic differences in biomarkers.

Over the last few years, newer anti-proteinuric agents and immunomodulatory drugs have either been approved by the FDA or are in the late phases of clinical trials for various proteinuric kidney diseases. The results of the STOP-IgAN and the recent TESTING trial have shown that the short-term beneficial effects of steroids on proteinuria and eGFR slope at six months wane over time, and there is a need for effective longer-term agents. The KDIGO guidelines development body on glomerular diseases has actively advocated enrolling patients prospectively in 'Clinical Trials'.

Platform trials are Multi-Arm and Multi-Stage (MAMS) randomised CTs comparing multiple parallel interventional groups against standardised common control groups with central coordination. It allows new interventions to be added, the control group to be updated throughout the trial, and the use of prespecified interim analysis plans for statistical efficiencies. Interventional groups can be introduced after the trial has started based on pre-specified criteria, and futile interventions may be stopped based on pre-specified interim analyses and trial-stopping rules.

This is a randomised controlled single-blind (outcome assessor) Platform trial, Multi-Arm and Multi-Stage. There is a single overarching protocol called a Master protocol. The master protocol, the common concurrent control arm for multiple interventions,the within-trial adaptations, the pre-specified interim analyses, and the pragmatic nature ensure greater acceptability and allow key trial characteristics to evolve. The overall strategy of the study relies strongly on pragmatic 'real world clinical situations' faced by practising nephrologists when treating adult patients with kidney biopsy-proven primary IgAN in South Asia. It will establish the 'GRACE Clinical Trial Network'.

The overarching trial hypothesis is that commonly available and approved generic drugs (low-dose oral prednisolone, gut-directed budesonide, mycophenolate mofetil, and hydroxychloroquine) in addition to Standard of Care (SoC), which is the maximal labelled or tolerated dose of renin-angiotensin system blockers (ACEi/ ARB) and a steady dose of sodium-glucose cotransporter 2 inhibitors (SGLT2i) can significantly improve the kidney outcomes at two years when compared to Standard of Care (SoC) alone in South Asian kidney biopsy-proven adult (≥18 years) primary IgAN who on follow-up remain at high risk of progression defined as UPCR ≥0.75g/g and baseline eGFR ≥20ml/min/1.73m2 despite good BP control. SoC is defined as a maximal labelled or tolerated dose of ACEi/ ARB and a steady dose of SGLT2i with a goal BP <140/90 mmHg for at least three months.

ELIGIBILITY:
Inclusion Criteria:

1. Must be able to provide a written informed consent form, which must be obtained before the initiation of study assessments.
2. Adults between 18-65 years of age.
3. Males or Females.
4. Diagnosis of primary IgAN as demonstrated by renal biopsy of any vintage if eGFR ≥45 mL/min/1.73 m2 or within the last ten years if eGFR <45 mL/min/1.73 m2. If diabetic, the biopsy vintage should be less than five years.
5. eGFR ≥20 mL/min/1.73 m2 at screening, as per the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation.
6. Total urine protein excretion ≥1 g per 24-hour or UPCR ≥ 0.75 g/g from an adequately measured 24-hour urine sample (24HUP) during the Screening Period.
7. Patient on the maximum labelled or tolerated dose of ACEi or ARB AND 10mg/d of Dapagliflozin (SGLT2i) for at least 12 weeks at screening and from screening to study Day 1.
8. Systolic blood pressure ≤140 mmHg and diastolic blood pressure ≤90 mmHg at randomisation. Other anti-hypertensives can be optimised during the screening period to achieve the BP goal.
9. A female is eligible if she is not pregnant and consents to avoid pregnancy during the study duration.

Exclusion Criteria:

1. IgAN secondary to another condition (e.g., liver cirrhosis) or other causes of mesangial IgA deposition such as systemic lupus erythematosus (SLE), dermatitis herpetiformis, ankylosing spondylitis, etc. IgA vasculitis (i.e., Henoch-Schonlein purpura) with biopsy-proven mesangial IgA deposition and no active skin vasculitis for the last year can be included.
2. Evidence of nephrotic syndrome at screening (serum albumin <3g/dL AND UPCR >3.5 g/g).
3. Evidence of rapidly progressive glomerulonephritis defined as loss of ≥ 50% of eGFR in three months before screening.
4. Concomitant kidney disease in addition to IgAN in kidney biopsy (e.g., diabetic nephropathy, primary focal segmental glomerulosclerosis, membranous nephropathy, C3 glomerulopathy, lupus nephritis).
5. Female patients planning pregnancy.
6. Concomitant co-morbidities like systemic autoimmune disorders, chronic active infections like tuberculosis, hepatitis B, hepatitis C and human immunodeficiency virus infection, chronic liver disease, and chronic obstructive pulmonary disease.
7. Renal or other organ transplantation before, or expected during, the study, except for corneal transplants.
8. Morbid obesity defined as BMI ≥ 40 kg/m2 at screening.
9. Uncontrolled diabetes as defined by HbA1c > 8% at screening.
10. History or diagnosis of demyelinating diseases such as multiple sclerosis or optic neuritis.
11. Prohibited medications:

    * Participants who received oral steroids over two weeks within 12 weeks before screening.
    * Immunosuppressive medications (e.g., MMF, azathioprine, cyclophosphamide, hydroxychloroquine) for treating IgAN within 12 weeks before screening.
    * Use of B-cell-directed biologic therapies, including belimumab, rituximab, and ocrelizumab, within six months before screening.
    * Use of other biologics (e.g., anti-TNF, abatacept, anti-IL-6) and investigational biologics within the last four weeks or five half-lives, whichever is longer, before the screening.
    * Use of traditional medications and/or Ayurvedic medications within 12 weeks before screening.
    * Use of endothelin receptor antagonists/ oral spironolactone or oral finerenone/ GLP-1 agonists/ hydroxychloroquine within 12 weeks before screening.
12. Patients with a history of unstable angina, Class III and IV congestive heart failure, and clinically significant arrhythmia, as judged by the Investigator.
13. Active clinically significant viral, bacterial, or fungal infection or any major episode of infection requiring hospitalisation or treatment with parenteral anti-infectives within four weeks before or during the Screening Visit.
14. History of malignancy within the past five years before Screening (except for adequately treated basal cell carcinoma or non-metastatic squamous cell carcinoma of the skin or cervical carcinoma in situ, with no evidence of recurrence).
15. Known hypersensitivity to any of the interventions.
16. Major surgery within six weeks before the Screening Visit.
17. Clinically significant history of alcohol or drug abuse in the one year before the Screening Visit as per the Investigator's opinion.
18. Unwillingness or lack of capacity to follow all study procedures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 585 (Estimated)
Dates: Start 2025-02-15 (Actual); Primary Completion 2029-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
To evaluate the mean change in annualized eGFR slope (ml/min/1.73m2) in the interventional and the active comparator arms. | Baseline, 3, 6, 9, 12, 15, 18 and 24 months
  Mean change in eGFR slope in ml/min/1.73m2/year

SECONDARY OUTCOMES:
To evaluate the mean change in UPCR ratio in the interventional and the active comparator arms. | Baseline, 6, 12, 18 and 24 months
  Mean change in Urine protein creatinine ratio in g/g. The mean change in UPCR ratio at 12 months is a pre-planned interim analysis for lack-of-benefit.
To evaluate the mean change in time averaged proteinuria in the interventional and the active comparator arms. | Baseline, 6, 12, 18 and 24 months
  Mean change in Time-averaged urine protein creatinine ratio in g/g
Proportion of participants reaching the composite endpoint | From enrollment to the end of treatment at 24 months
  Composite end-point is defined as ≥50% decline in eGFR sustained for at least 28 days, end-stage kidney disease requiring renal replacement therapy, or death.
Proportion of participants having rapidly progressive kidney disease | From enrollment to the end of treatment at 24 months
  Rapidly progressive kidney disease is defined as ≥50% decline in eGFR over three months
Proportion of participants reaching eGFR <15 ml/min/1.73 m2 | From enrollment to the end of treatment at 24 months
  <15ml/min/1.73m2 eGFR sustained for at least 28 days
Proportion of participants' using rescue medication | From enrollment to the end of treatment at 24 months
  Using of other immunomodulatory treatments after ≥50% decline in eGFR over three months
Adverse Events | From enrollment to the end of treatment at 24 months
  Percentage adverse events in clinical and laboratory tests.
Glucocorticoid Toxicity Index | Baseline, 6months, 12 months
  Change in Glucocorticoid Toxicity Index (GTI) score for prednisolone and budesonide arms.
Medication Adherence | From enrollment to the end of treatment at 24 months
  To evaluate the proportion of participants with Medication Adherence in the interventional and the active comparator arms.
To evaluate participant related outcome measure (PROM) by EQ-5D-5L | Baseline, 12 and 24 months
  EQ-5D-5L study instrument
To evaluate PROM by KDQOL-36 | Baseline, 12 and 24 months
  KDQOL-36 study instrument
To evaluate PROM py FACIT-F | Baseline, 12 and 24 months
  FACIT-F study instrument

OTHER OUTCOMES:
Serum biomarker profile | Baseline, 12, 24 months
  To evaluate the longitudinal change in serum biomarker profile from baseline to two years. This is an exploratory objective and the bio samples will be stored and the evaluation done later with supplemental funds.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Barratt, PhD, FRCP, Study Chair — University of Leicester; George T John, DM, FRCP, FRACP, Study Chair — Royal Brisbane and Women's Hospital
Locations (12):
- India (12):
  - Muljibhai Patel Urological Hospital, Nadiād, Gujarat
  - JSS Medical College, Mysuru, Karnataka
  - Kasturba Medical College, Manipal, Udupi, Karnataka
  - KEM Hospital, Mumbai, Maharashtra
  - Safdarjung Hospital, Ansari Nagar East, Delhi, New Delhi
  - AIIMS Bhubaneswar, Bhubaneswar, Odisha
  - JIPMER, JIPMER Campus, Puducherry, Puducherry
  - Madras Medical College, Chennai, Tamil Nadu
  - Christian Medical College Vellore, Vellore, Tamil Nadu
  - Nizams Institute of Medical Sciences, Hyderabad, Telangana
  - Osmania Medical College, Hyderabad, Telangana
  - Sanjay Gandhi Post Graduate Institute of Medical Sciences, Lucknow, Uttar Pradesh

IPD SHARING:
Plan to Share IPD: Yes
All de-identified individual-level data, as permitted by the local law, will be made available on Mendeley Data. Access to data will be possible by writing to gracetrials@cmcvellore.ac.in or suceena@cmcvellore.ac.in on or after 31 Dec 2030.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within 6 months of data lock at the end of the trial and for a period of five years thereafter.
Access Criteria: Upon providing a draft hypothesis and analysis plan.
URL: https://gracetrials.cmcv.ac.in/